CLINICAL TRIAL: NCT01817335
Title: Pilot Study of Psycho-Educational Group for Young Adults (YA) on Treatment: Impact on Knowledge, Distress, and Satisfaction
Brief Title: Psycho-Educational Program in Increasing Knowledge and Satisfaction and Decreasing Distress in Younger Patients With Cancer Receiving Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13128; NCI-2013-00589 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-19; First posted 2013-03-25 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Malignant Neoplasm; Psychosocial Effects of Cancer and Its Treatment
MeSH Terms: conditions — Neoplasms | interventions — Psychiatric Rehabilitation; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (psycho-educational program) (Experimental): Patients participate in a psycho-educational program focused on medical/symptom management and communication with a medical team, coping skills, self image, and relationships and communication for 1.5 hours once weekly for 6 weeks.
  Interventions: Procedure: psychosocial assessment and care; Other: educational intervention; Other: communication skills training; Other: questionnaire administration

INTERVENTIONS:
Procedure: psychosocial assessment and care — Participate in psycho-educational program
  Other Names: psychosocial assessment; psychosocial assessment/care; psychosocial care; psychosocial care/assessment; psychosocial studies
Other: educational intervention — Participate in psycho-educational program
  Other Names: intervention, educational
Other: communication skills training — Participate in psycho-educational program
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies psycho-educational program in increasing knowledge and satisfaction and decreasing distress in younger patients with cancer receiving treatment. Psycho-educational program may increase knowledge and satisfaction and decrease distress in younger patients with cancer receiving treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Providing a psycho-educational group to young adults while examining the feasibility of such a group with patients on treatment.

II. Examining effectiveness of the program through evaluating pre-post changes in participant distress, evaluating increases in participant' knowledge regarding disease issues and coping, and evaluating participant satisfaction.

OUTLINE:

Patients undergo psycho-educational program comprising medical/symptom management and communication with a medical team, coping skills, self image, and relationships and communication for 1.5 hours once weekly for 6 weeks.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Currently in active treatment (diagnosed and receiving treatment within 2 weeks of initial study enrollment; active treatment includes currently receiving any of the following: chemotherapy, radiation therapy, maintenance drugs, surgery, clinical trial enrollment, or current relapse/secondary malignancy)
* Inpatient or outpatient
* Cancer diagnosis
* Physician approval
* Informed consent

Exclusion Criteria:

* Significant psychiatric or developmental issues, as determined by screening interview conducted by psychologist or clinical social worker
* Currently off treatment (longer than 2 weeks at the time of enrollment)
* In isolation or with isolation precautions
* Non-English speaking

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who are unable to attend all the sessions | Up to 30 days

SECONDARY OUTCOMES:
Mean of the YA (Young Adult) Patient Satisfaction evaluations | Up to 30 days
  A questionnaire was developed to measure participant satisfaction with the format and material of the psycho-educational program. Satisfaction measures will be provided for completion at the end of sessions 2 through 5 and 30 days post intervention. Changes in the mean of the Questionnaire responses will be analyzed using a paired t-test and calculations of simple frequency and descriptive statistics will be used to summarize the data and program evaluations.
Mean of the Pre/Post Test Knowledge Questionnaire | Up to 30 days
  A questionnaire was developed based on the psycho-educational material to assess increases in knowledge and retention. The questionnaire will be administered pre-intervention and 30 days post-intervention. Additionally, relevant items from the questionnaire will be administered at the end of the relevant educational session. For instance, self image questions from the questionnaire will be administered at the end of the self-image session in addition to the pre and post administration of the entire questionnaire. Changes in the mean of the Questionnaire responses will be analyzed using a paired t-test and calculations of simple frequency and descriptive statistics will be used to summarize the data and program evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanelle Folbrecht, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States